CLINICAL TRIAL: NCT01920568
Title: DCA114273: A Study Comparing Denosumab With Zoledronic Acid in Subjects of Asian Ancestry With Bone Metastases From Solid Tumors
Brief Title: A Study to Compare Denosumab With Zoledronic Acid in Subjects With Bone Metastases From Solid Tumors
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 114273
Record Dates: First submitted 2013-08-08; First posted 2013-08-12 (Estimated); Results first posted 2016-08-25 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2016-07

CONDITIONS: Fractures, Bone
Keywords: GSK2371746; Denosumab; China; skeletal-related events; bone metastases; bridging study; solid tumors
MeSH Terms: conditions — Fractures, Bone | interventions — Denosumab; Zoledronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Denosumab 120 mg (Experimental): Subjects will be administered with Denosumab 120 mg subcutaneous (SC) injection for a maximum of 13 doses and placebo IV infusion over >=15 minutes once every 4 weeks.
  Interventions: Biological: Denosumab 70 mg/mL; Drug: Placebo IV; Dietary Supplement: Calcium supplement; Dietary Supplement: Vitamin D supplement
- Zoledronic acid 4 mg (Experimental): Subjects will be administered with Zoledronic acid 4 mg IV infusion over a minimum of 15 minutes for a maximum of 13 doses and placebo SC once every 4 weeks.
  Interventions: Drug: Zoledronic acid 4 mg; Drug: Placebo SC; Dietary Supplement: Calcium supplement; Dietary Supplement: Vitamin D supplement

INTERVENTIONS:
Biological: Denosumab 70 mg/mL — Denosumab will be given as a SC injection of 120 mg by administering a 1.7 mL volume in a single injection
  Arms: Denosumab 120 mg
Drug: Zoledronic acid 4 mg — Zoledronic acid 4 mg (or equivalent clearance-adjusted dose in subjects with baseline creatinine clearance <=60 ml/min) will be diluted in either 0.9% sodium chloride or 5% dextrose injection and administered IV.
  Arms: Zoledronic acid 4 mg
Drug: Placebo IV — The placebo will consist of 1.7 mL 0.9% w/v sodium chloride
  Arms: Denosumab 120 mg
Drug: Placebo SC — The placebo will consist of either 0.9% w/v sodium chloride or 5% dextrose injection
  Arms: Zoledronic acid 4 mg
Dietary Supplement: Calcium supplement — Subjects are strongly recommended to take daily supplements of at least 500 mg calcium from the day of consent and until completion of the Week 73 follow-up visit.
Dietary Supplement: Vitamin D supplement — Subjects are strongly recommended to take daily supplements of at least 400 IU of vitamin D from the day of consent and until completion of the Week 73 follow-up visit.

SUMMARY:
This is a randomized, double-blind, double-dummy study designed to provide bridging data in an Asian population to Amgen's studies of denosumab in subjects with bone metastases from solid tumors. The study is designed to provide data to a large global dataset of phase-III studies including breast cancer, prostate cancer, and all solid tumors, plus multiple myeloma, to support the regulatory approval for marketing and patient access to denosumab for the prevention of SREs in Chinese subjects with bone metastases from solid tumors. The primary objective of this study is to evaluate and compare the percent change from baseline to Week 13 in the bone marker urinary amino-terminal cross-linking telopeptide of type I collagen (uNTx) corrected for urine creatinine (uNTx/uCr) in subjects treated with denosumab to those treated with zoledronic acid. The study is designed to test the superiority of denosumab over zoledronic acid.

ELIGIBILITY:
Inclusion Criteria:

* Subject understands the nature and purpose of this study and the study procedures, which have been explained by the Investigator or delegate, and subject has signed the written informed consent for the overall study. The subject must sign a separate written informed consent to be eligible for enrolment in the pharmacokinetic substudy.
* Adult (aged >=18 years) of Asian ancestry with a histologically or cytologically confirmed solid tumor. In addition, subjects who are enrolled at a center in mainland China or at an SFDA-certified center in Hong Kong including the approximately 33 subjects in the pharmacokinetic substudy must be of Chinese race, ancestry, or heritage. Subjects enrolled in other regions or countries, such as Taiwan and Singapore, or at a non-SFDA-certified center in Hong Kong, are not required to be of Chinese race or ancestry.
* Current or prior documented radiographic evidence (i.e., x-ray, computer tomography [CT], or magnetic resonance imaging [MRI]) of at least 1 bone metastasis.
* Female subjects of childbearing potential must have a negative serum or urine pregnancy test within 7 days of first dose of study treatment and agree to use effective contraception, as defined below, during the study and for 6 months after end of study treatment. Women who report having a pregnancy during this study will be followed for birth outcomes. GSK acceptable contraceptive methods, when used consistently and in accordance with both the product label and the instructions of the physician, are as follows: An intrauterine device or intrauterine system with a documented failure rate of less than 1% per year; Male partner sterilization prior to the female subject's enrollment and the male is the sole sexual partner for that subject; the information on the male sterility can come from the site personnel's review of subject's medical records; medical examination of the subject and/or semen analysis; or interview with the subject on his medical history; complete abstinence from sexual intercourse for 14 days prior to first dose of study treatment, through the dosing period, and for at least 7 months after the last dose of study treatment; double-barrier contraception: male condom combined with a female diaphragm, either with or without a vaginal spermicide (foam, gel, film, cream, or suppository); implants of levonorgestrel or etonogestrel where not contraindicated for this patient population or per local practice; injectable progesterone where not contraindicated for this patient population or per local practice; percutaneous contraceptive patches where not contraindicated for this patient population or per local practice; Oral contraceptives (either combined or progesterone only) where not contraindicated for this patient population or per local practice. Females of child bearing potential who do not have male partners as part of their preferred and usual lifestyle are not required to use contraception.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2 (refer protocol for details).
* Adequate baseline organ function as defined by the following criteria: Serum aspartate aminotransferase (AST) <=2.0 x upper limit of normal (ULN); Serum alanine aminotransferase (ALT) <=2.0 x ULN; Serum total bilirubin <=1.0 x ULN; creatinine clearance (calculated using the Cockcroft-Gault formula) >=30 milliliter per minute (mL/min); serum calcium or albumin-adjusted serum calcium >=2.0 millimole per liter (mmol/L) (8.0 mg/dL) and <=2.9 mmol/L (11.5 miligram per deciliter [mg/dL]). Subjects must not have taken supplemental calcium for at least 8 hours prior to collection of the blood sample for screening serum calcium determination.
* Life expectancy of at least 6 months, in the opinion of the Investigator.

Exclusion Criteria:

* Any serious and/or unstable pre-existing medical, psychiatric disorder, or other conditions that, in the opinion of the Investigator, could interfere with subject's safety, obtaining informed consent or compliance to the study procedures; The Investigator should consult the GSK Medical Monitor prior to enrolling a subject if s/he is unsure if a condition might interfere with the subject's safety or participation in this study.
* Any prior treatment with intravenous (IV) or oral bisphosphonates.
* Prior treatment with denosumab.
* Planned radiation therapy or surgery to bone.
* Known brain metastases.
* Prior history or current evidence of osteomyelitis or osteonecrosis of the jaws (ONJ), an active dental or jaw condition that requires oral surgery, non-healed dental or oral surgery, or planned invasive dental procedure over the course of the study.
* Evidence of any of the following conditions per subject self report or medical chart review: any prior or current malignancy (other than the cancer under study in this protocol) with active disease within 3 years before randomization; unstable liver disease (as defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, or persistent jaundice), known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones); known infection with human immunodeficiency virus (HIV); active infection with hepatitis B or hepatitis C virus.
* Pregnant women, women planning to become pregnant within 7 months after end of study treatment, and women who are breastfeeding. Women who are breast feeding should discontinue nursing prior to the first dose of study treatment and should refrain from nursing throughout the treatment period and for 7 months following their last dose of study treatment.
* Male subjects unable or unwilling to use adequate contraception methods during the study and for 6 months after end of study treatment should be excluded.
* Subject is currently enrolled in another investigational device or investigational product study, or has not completed at least 30 days, 5 half lives, or the duration of biological effect, whichever is longer, since ending such a study.
* Known sensitivity to any of the investigational products or supplements to be administered during the study (i.e., zoledronic acid, mammalian derived products, calcium, or vitamin D).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 487 (Actual)
Dates: Start 2013-08; Primary Completion 2015-02 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (15):
- China (12):
  - GSK Investigational Site, Guangzhou, Guangdong
  - GSK Investigational Site, Wuhan, Hubei
  - GSK Investigational Site, Nanjing, Jiangsu
  - GSK Investigational Site, Changchun, Jilin
  - GSK Investigational Site, Chengdu, Sichuan
  - GSK Investigational Site, Hangzhou, Zhejiang
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Fuzhou
  - GSK Investigational Site, Hangzhou
  - GSK Investigational Site, Harbin
  - GSK Investigational Site, Shanghai
  - GSK Investigational Site, Tianjin
- GSK Investigational Site, Singapore, Singapore
- Taiwan (2):
  - GSK Investigational Site, Taichung
  - GSK Investigational Site, Taoyuan District

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study consisted of three phases: Screening period , 49-week Double-blind treatment period and Follow-up period. The total participation time in the study was approximately 77 weeks.
Pre-assignment Details: A total of 487 participants (par.) were randomized in a 2:1 ratio to receive one of the two study treatments. A total of 485 participants received at least single dose of investigational products (IP).
Groups:
- Denosumab 120 mg: Participants received denosumab 120 milligrams (mg) as subcutaneous (SC) injection for a maximum of 13 doses and placebo as intravenous (IV) infusion over a minimum of 15 minutes once every 4 weeks up to 49 weeks. Participants also received daily oral supplementation of >= 500 mg elemental calcium and >=400 international unit (IU) of vitamin D.
- Zoledronic Acid 4 mg: Participants received zoledronic acid 4 mg as IV infusion over a minimum of 15 minutes for a maximum of 13 doses and placebo as SC once every 4 weeks up to 49 weeks. Participants also received daily oral supplementation of >= 500 mg elemental calcium and >=400 IU of vitamin D.
Period: Overall Study
Arm/Group | Denosumab 120 mg | Zoledronic Acid 4 mg
Started | 326 | 159
Completed | 175 | 75
Not Completed | 151 | 84
Not completed — Adverse Event | 27 | 8
Not completed — Protocol Violation | 5 | 3
Not completed — Lost to Follow-up | 2 | 2
Not completed — Physician Decision | 13 | 4
Not completed — Withdrawal by Subject | 79 | 55
Not completed — Death due to disease progression | 25 | 12

BASELINE CHARACTERISTICS:
Groups:
- Denosumab 120 mg: Participants received denosumab 120 mg as SC injection for a maximum of 13 doses and placebo as IV infusion over a minimum of 15 minutes once every 4 weeks up to 49 weeks. Participants also received daily oral supplementation of >= 500 mg elemental calcium and >=400 IU of vitamin D.
- Total: Total of all reporting groups
Arm/Group | Denosumab 120 mg | Zoledronic Acid 4 mg | Total
Number analyzed (Participants) | 326 | 159 | 485
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.0 (11.36) | 53.6 (11.45) | 53.9 (11.38)
Gender [Count of Participants; unit: Participants]
  Female | 222 | 105 | 327
  Male | 104 | 54 | 158
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian - East Asian Heritage | 312 | 158 | 470
  Asian - South East Asian Heritage | 14 | 1 | 15

OUTCOME MEASURES:

1. Primary Outcome: Percent Change (Chg) From Baseline (BL) to Week (Wk)13 in Urinary Amino-terminal Cross-linking Telopeptide of Type I Collagen Corrected for Urine Creatinine (uNTx/uCr)
Description: uNTx/uCr is the bone turnover marker correlated with the presence and extent of metastases, and the prognosis and response to bone targeted treatment (trt). uNTx/uCr was expressed in nanomoles bone collagen equivalent per millimole (nM BCE/mM). Primary objective: to compare the effect of denosumab with that of zoledronic acid on % chg from BL in uNTx/uCr at Wk 13 in par. of Asian ancestry with bone metastases from solid tumors. BL value is the most recent, non-missing value prior to or on the 1st study trt dose date. Chg from BL is the value at Wk13 minus BL value. Percent chg from BL is the chg from BL / BL value * 100. For missing Wk 13 observations, the last post-BL value was carried forward to obtain the Wk 13 value.
Time Frame: Baseline (BL) and Week (Wk) 13
Population: Full-Analysis-Set Intent-to-Treat (FAS-ITT) Population: comprised of all randomized participants regardless of whether or not study treatment was administered. Only those participants with values at Baseline and Week 13 were included in the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Denosumab 120 mg | Zoledronic Acid 4 mg
Number analyzed (Participants) | 322 | 154
Percent change | -81.9 [-83.1 to -80.6] | -75.2 [-77.6 to -72.5]
Statistical Analysis 1: Comparison: Denosumab 120 mg vs Zoledronic Acid 4 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.316, 95% CI 2-sided [-0.440 to -0.192] — Primary analysis evaluated the log transformed chg from BL, i.e. log[(Wk 13 uNTx/Cr) / (BL uNTx/Cr)] by ANCOVA model with trt group as main effect and the stratification factor (breast cancer, yes or no) and log transformed BL value as covariates

2. Secondary Outcome: Percentage Change From Baseline to Week 13 in Urinary Amino-terminal Cross-linking Telopeptide of Type I Collagen of Type I Collagen Corrected for Urine Creatinine (uNTx/uCr) in Chinese Participants.
Description: uNTx/uCr is the bone turnover marker correlated with the presence and extent of metastases, and the prognosis and response to bone targeted treatment. uNTx/uCr was expressed in nanomoles bone collagen equivalent per millimole (nM BCE/mM). Secondary objective: to compare the effect of denosumab with that of zoledronic acid on % chg from BL in uNTx/uCr at Wk 13 in par. of Chinese ancestry with bone metastases from solid tumors. Baseline value is the most recent, non-missing value prior to or on the first study treatment dose date. Change from Baseline is the value at Week 13 minus Baseline value. Percent chg from BL is the chg from BL / BL value * 100. For missing Wk 13 observations, the last post-BL value was carried forward to obtain the Wk 13 value.
Time Frame: Baseline and Week 13
Population: FAS-ITT Population. Chinese participants.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Denosumab 120 mg | Zoledronic Acid 4 mg
Number analyzed (Participants) | 296 | 147
Percent change | -82.2 [-83.4 to -80.8] | -75.6 [-78.0 to -72.9]
Statistical Analysis 1: Comparison: Denosumab 120 mg vs Zoledronic Acid 4 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.316, 95% CI 2-sided [-0.444 to -0.188] — Secondary analysis evaluated the log transformed chg from BL, ie log[(Wk 13 uNTx/Cr)/(BL uNTx/Cr)] by ANCOVA model with trt group as main effect and the stratification factor (Chinese participants, yes or no) and log transformed BL value

3. Secondary Outcome: Percentage Change From Baseline to Week 13 in Urinary Amino-terminal Cross-linking Telopeptide of Type I Collagen of Type I Collagen Corrected for Urine Creatinine (uNTx/uCr) in Participants With Advanced Breast Cancer.
Description: uNTx/uCr is the bone turnover marker correlated with the presence and extent of metastases, and the prognosis and response to bone targeted treatment. uNTx/uCr was expressed in nanomoles bone collagen equivalent per millimole (nM BCE/mM). Secondary objective: to compare the effect of denosumab with that of zoledronic acid on % chg from BL in uNTx/uCr at Wk 13 in breast cancer par. with bone metastases from solid tumors. Baseline value is the most recent, non-missing value prior to or on the first study treatment dose date. Change from Baseline is the value at Week 13 minus Baseline value. Percent chg from BL is the chg from BL / BL value * 100. For missing Wk 13 observations, the last post-BL value was carried forward to obtain the Wk 13 value.
Time Frame: Baseline and Week 13
Population: FAS-ITT Population. Participants with advanced breast cancer.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Denosumab 120 mg | Zoledronic Acid 4 mg
Number analyzed (Participants) | 160 | 77
Percent change | -80.9 [-82.7 to -78.9] | -72.4 [-76.1 to -68.2]
Statistical Analysis 1: Comparison: Denosumab 120 mg vs Zoledronic Acid 4 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.366, 95% CI 2-sided [-0.539 to -0.193] — Secondary analysis evaluated the log transformed chg from BL, i.e. log[(Wk 13 uNTx/Cr) / (BL uNTx/Cr)] by ANCOVA model with trt group as main effect, stratification factor (Breast cancer, yes or no) and log transformed BL value as covariates

4. Secondary Outcome: Percent Change From Baseline in the Serum Bone-specific Alkaline Phosphatase (s-BALP) at Week 13.
Description: Baseline value is the most recent, non-missing value prior to or on the first study treatment dose date. Change from Baseline is the value at Indicated visit minus Baseline value. Percent change from Baseline is the change from Baseline divided by Baseline value multiplied by 100.
Time Frame: Baseline and Week 13
Population: FAS-ITT Population. All participants who were randomized and had a observed values at Baseline and Week 13 were used in the analysis.
Measure: Median (Full Range); unit: Percent change
Arm/Group | Denosumab 120 mg | Zoledronic Acid 4 mg
Number analyzed (Participants) | 294 | 134
Percent change | -36.8 [-96.2 to 93.8] | -30.3 [-91.7 to 345.9]

5. Secondary Outcome: Number of Participants With Any Adverse Events (AEs), Serious Adverse Events (Non-fatal Serious Adverse Events and Fatal Serious Adverse Events)
Description: An AE is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. A serious adverse event (SAE) is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect or other events that may jeopardize the participant or may require medical or surgical intervention to prevent one of the outcome listed above, liver injury and impaired liver function and grade 4 laboratory abnormalities. Number of participants with any AEs, non-fatal SAEs, fatal SAEs have been presented.
Time Frame: From start of IP through the Study Phase (49 weeks post-dose) (assessed up to 73 weeks)
Population: Full-Analysis-Set Safety (FAS-Safety) Population: comprised of all randomized participants who received at least one dose of study treatment and was based on the actual study treatment received (if this differed from that to which the participant was randomized).
Measure: Number; unit: Participants
Arm/Group | Denosumab 120 mg | Zoledronic Acid 4 mg
Number analyzed (Participants) | 326 | 159
Participants
  Any AEs | 291 | 145
  Any SAEs | 46 | 14
  Any Fatal SAEs | 25 | 7
  Any Non-Fatal SAEs | 25 | 7

6. Secondary Outcome: Number of Participants With Worst-case (WC) On-therapy Increase in the Indicated Clinical Chemistry Parameters From Baseline Grade to the Indicated Grade.
Description: Clinical chemistry parameters were measured at the Screening and Weeks 2, 5, 9, 13, 25, 37, and 53 visits. Clinical chemistry parameters measured on-study included albumin, alkaline phosphatase (ALP), alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin, calcium (Ca), creatinine, magnesium, and phosphorous (P) inorganic. All reported values are of participants with worst-case on-therapy increase to the specified grade: Any increase, that is, worst-case increase to grade 1, 2, 3, or 4 (any grade); worst-case increase to grade 3 (WC G3); and worst-case increase to grade 4 (WC G4). The National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) was used for grading. Participants with missing Baseline grade were assumed to have a Baseline grade of 0. The worst-case during the on-therapy period was determined taking into account both scheduled and unscheduled assessments.
Time Frame: Baseline and up to last study-related visit (up to 53 weeks)
Population: FAS-Safety Population. Only participants whose indicated on-therapy laboratory values were available (represented by n=X, X in the category title) were analyzed.
Measure: Number; unit: Participants
Arm/Group | Denosumab 120 mg | Zoledronic Acid 4 mg
Number analyzed (Participants) | 326 | 159
Participants
  Albumin (hyperalbuminemia), any grade, n=324, 156 | 0 | 0
  Albumin (hyperalbuminemia), WC G3, n=324, 156 | 0 | 0
  Albumin (hyperalbuminemia), WC G4, n=324, 156 | 0 | 0
  Albumin (hypoalbuminemia), any grade, n=324, 156 | 45 | 26
  Albumin (hypoalbuminemia), WC G3, n=324, 156 | 1 | 0
  Albumin (hypoalbuminemia), WC G4, n=324, 156 | 0 | 0
  ALP, any grade, n=324, 156 | 67 | 31
  ALP, WC G3, n=324, 156 | 7 | 2
  ALP, WC G4, n=324, 156 | 0 | 0
  ALT, any grade, n=324, 156 | 137 | 59
  ALT, WC G3, n=324, 156 | 7 | 4
  ALT, WC G4, n=324, 156 | 0 | 0
  AST, any grade, n=323, 155 | 117 | 61
  AST, WC G3, n=323, 155 | 7 | 4
  AST, WC G4, n=323, 155 | 0 | 0
  Total Bilirubin, any grade, n=324, 155 | 34 | 16
  Total Bilirubin, WC G3, n=324, 155 | 2 | 0
  Total Bilirubin, WC G4, n=324, 155 | 2 | 1
  Calcium (hypercalcemia), any grade, n=324, 156 | 4 | 3
  Calcium (hypercalcemia), WC G3, n=324, 156 | 0 | 0
  Calcium (hypercalcemia), WC G4, n=324, 156 | 0 | 1
  Calcium (hypocalcemia), any grade, n=324,156 | 78 | 28
  Calcium (hypocalcemia), WC G3, n=324, 156 | 5 | 0
  Calcium (hypocalcemia), WC G4, n=324, 156 | 1 | 0
  Creatinine, any grade, n=324, 156 | 16 | 13
  Creatinine, WC G3, n=324, 156 | 1 | 0
  Creatinine, WC G4, n=324, 156 | 0 | 0
  Magnesium (hypermagnesemia), any grade, n=324, 156 | 4 | 0
  Magnesium (hypermagnesemia), WC G3, n=324, 156 | 2 | 0
  Magnesium (hypermagnesemia), WC G4, n=324, 156 | 0 | 0
  Magnesium (hypomagnesemia), any grade, n=324, 156 | 8 | 2
  Magnesium (hypomagnesemia), WC G3, n=324, 156 | 0 | 0
  Magnesium (hypomagnesemia), WC G4, n=324, 156 | 0 | 0
  P,inorganic(hyperphosphatemia),any grade,n=323,156 | 0 | 0
  P, inorganic (hyperphosphatemia),WC G3, n=323, 156 | 0 | 0
  P, inorganic (hyperphosphatemia),WC G4, n=323, 156 | 0 | 0
  P,inorganic(hypophosphatemia),any grade,n=323, 156 | 124 | 35
  P, inorganic (hypophosphatemia),WC G3, n=323, 156 | 35 | 9
  P, inorganic (hypophosphatemia), WC G4, n=323, 156 | 1 | 0

7. Secondary Outcome: Number of Participants With Worst-case On-therapy Increase in the Indicated Hematology Parameters From Baseline Grade to the Indicated Grade.
Description: Hematology parameters included hemoglobin, lymphocytes, platelet count, total neutrophils, white blood cell (WBC) count. All reported values are of participants with worst-case on-therapy increase to the specified grade: Any increase, that is, worst-case increase to grade 1, 2, 3, or 4 (any grade); worst-case increase to grade 3 (WC G3); and worst-case increase to grade 4 (WC G4). Participants with missing Baseline grade were assumed to have a Baseline grade of 0. The worst-case during the on-therapy period was determined taking into account both scheduled and unscheduled assessments.
Time Frame: Baseline and up to last study-related visit (up to 53 weeks)
Population: FAS-Safety Population. Only participants whose indicated on-therapy lab values were available (represented by n=X, X in the category titles) were analyzed.
Measure: Number; unit: Participants
Arm/Group | Denosumab 120 mg | Zoledronic Acid 4 mg
Number analyzed (Participants) | 326 | 159
Participants
  Hemoglobin, any grade, n=316, 147 | 139 | 69
  Hemoglobin, WC G3, n=316, 147 | 24 | 11
  Hemoglobin, WC G4, n=316, 147 | 0 | 0
  Lymphocyte count decreased, any grade, n=315, 147 | 77 | 47
  Lymphocyte count decreased, WC G3, n=315, 147 | 21 | 14
  Lymphocyte count decreased, WC G4, n=315, 147 | 1 | 1
  Lymphocyte count increased, any grade, n=315, 147 | 2 | 2
  Lymphocyte count increased, WC G3, n=315, 147 | 0 | 0
  Lymphocyte count increased, WC G4, n=315, 147 | 0 | 0
  Platelet count, any grade, n=314, 144 | 77 | 48
  Platelet count, WC G3, n=314, 144 | 2 | 5
  Platelet count, WC G4, n=314, 144 | 2 | 1
  Total neutrophils, any grade, n=315, 147 | 124 | 58
  Total neutrophils, WC G3, n=315, 147 | 40 | 19
  Total neutrophils, WC G4, n=315, 147 | 12 | 8
  WBC count, any grade, n=315, 147 | 138 | 78
  WBC count, WC G3, n=315, 147 | 25 | 19
  WBC count, WC G4, n=315, 147 | 2 | 1

8. Secondary Outcome: Number of Participants With Confirmed Anti-denosumab Antibody Formation at Day 1, Week 25 and Week 53.
Description: Anti-denosumab antibody formation was assessed at Day 1, Week 25 and Week 53. Binding antibody assay was used to assess number of participants with anti-denosumab antibody.
Time Frame: Day 1, Week 25 and Week 53
Population: FAS-Safety Population. Only those participants on whom anti-denosumab antibody formation was analyzed at specified time point is presented (represented by n=X, X in the category titles).
Measure: Number; unit: Participants
Arm/Group | Denosumab 120 mg | Zoledronic Acid 4 mg
Number analyzed (Participants) | 326 | 159
Participants
  Day 1, n = 326, 158 | 0 | 0
  Week 25, n = 256, 115 | 0 | 0
  Week 53, n = 180, 76 | 0 | 0

9. Secondary Outcome: Serum Concentration of Denosumab on Day 1, at Week 2, Week 5, Week 9, Week 13, Week 17, Week 19, Week 21, Week 25 and Week 49
Description: Blood samples were drawn on study Day 1, pre-dose; 4 hours, 24 hours, and at Week 2 (168 hours); then pre-dose at Week 5, Week 9, Week 13, Week 17, Week 19 (no dose), Week 21, Week 25, and Week 49.
Time Frame: Samples were collected at pre-dose (Day 1); 4 hours, 24 hours, 168 hours post-dose; pre-dose at Week 5, Week 9, Week 13, Week 17; Week 19 (at 336 hours); pre-dose at Week 21, Week 25, Week 49
Population: Pharmacokinetic (PK) Population: comprised of participants who signed informed consent to participate in the PK sub-study and who had their PK parameters evaluable according to GSK standards. Only those participants with evaluable parameters are included (represented by n=X in the category titles).
Measure: Geometric Mean (95% Confidence Interval); unit: micrograms per milliliter (µg/mL)
Groups:
- Denosumab 120 mg: Participants received denosumab 120 mg as SC injection for a maximum of 13 doses and placebo as IV infusion over a minimum of 15 minutes once every 4 weeks. Participants also received daily oral supplementation of >= 500 mg elemental calcium and >=400 IU of vitamin D.
Arm/Group | Denosumab 120 mg
Number analyzed (Participants) | 26
micrograms per milliliter (µg/mL)
  Day 1, Pre-dose, n=26 | 0 [0 to 0]
  Day 1, 4 hours post-dose, n=26 | 777.1 [574.2 to 1051.6]
  Day 1, 24 hours post-dose, n=26 | 5521.6 [4744.2 to 6426.3]
  Week 2, 168 hours post-dose, n=26 | 11701.1 [10554.0 to 12973.0]
  Week 5, Pre-dose, n=25 | 8658.1 [7631.1 to 9823.3]
  Week 9, Pre-dose, n=25 | 12086.4 [10284.9 to 14203.4]
  Week 13, Pre-dose, n=25 | 14867.5 [12515.5 to 17661.6]
  Week 17, Pre-dose, n=24 | 16543.3 [13871.8 to 19729.2]
  Week 19, 336 hours, n=22 | 20802.4 [16280.7 to 26579.9]
  Week 21, Predose, n=21 | 14508.0 [10907.0 to 19297.9]
  Week 25, Predose, n=22 | 16619.0 [13354.9 to 20681.0]
  Week 49, Predose, n=19 | 20029.2 [16282.7 to 24637.9]

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from start of IP through the Study Phase (49 weeks post-dose) (assessed up to 73 weeks).
Description: On-treatment SAEs and non-serious AEs are reported for the Safety Population, which comprises of all randomized participants who received at least one dose of study treatment and is based on the actual study treatment received (if this differs from that to which the participant was randomized).
Groups:
- Zoledronic Acid 4 mg: Participants received zoledronic acid 4 mg as IV infusion over a minimum of 15 minutes for a maximum of 13 doses and placebo as SC once every 4 weeks. Participants also received daily oral supplementation of >= 500 mg elemental calcium and >=400 IU of vitamin D.
Arm/Group | Denosumab 120 mg | Zoledronic Acid 4 mg
Serious Adverse Events (participants affected / at risk) | 46/326 | 14/159
Other Adverse Events (participants affected / at risk) | 268/326 | 136/159
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Denosumab 120 mg (N=326) | Zoledronic Acid 4 mg (N=159)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Pneumonia (Infections and infestations) | 3 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Disease progression (General disorders) | 3 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Death (General disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 2
Loss of consciousness (Nervous system disorders) | 2 | 0
Lung infection (Infections and infestations) | 2 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Sepsis (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Anal abscess (Infections and infestations) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Escherichia bacteraemia (Infections and infestations) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Gastroenteritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Liver injury (Hepatobiliary disorders) | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Streptococcal sepsis (Infections and infestations) | 0 | 1
Subdural hygroma (Nervous system disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0
Venous thrombosis (Vascular disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Denosumab 120 mg (N=326) | Zoledronic Acid 4 mg (N=159)
White blood cell count decreased (Investigations) | 68 | 38
Neutrophil count decreased (Investigations) | 55 | 30
Alanine aminotransferase increased (Investigations) | 56 | 28
Aspartate aminotransferase increased (Investigations) | 49 | 26
Platelet count decreased (Investigations) | 19 | 10
Weight decreased (Investigations) | 16 | 10
Anaemia (Blood and lymphatic system disorders) | 81 | 39
Leukopenia (Blood and lymphatic system disorders) | 55 | 27
Neutropenia (Blood and lymphatic system disorders) | 54 | 25
Thrombocytopenia (Blood and lymphatic system disorders) | 20 | 14
Bone marrow failure (Blood and lymphatic system disorders) | 17 | 8
Nausea (Gastrointestinal disorders) | 57 | 23
Constipation (Gastrointestinal disorders) | 34 | 23
Vomiting (Gastrointestinal disorders) | 30 | 15
Diarrhoea (Gastrointestinal disorders) | 19 | 15
Pyrexia (General disorders) | 41 | 32
Fatigue (General disorders) | 30 | 17
Asthenia (General disorders) | 23 | 10
Pain (General disorders) | 23 | 8
Decreased appetite (Metabolism and nutrition disorders) | 61 | 32
Hypocalcaemia (Metabolism and nutrition disorders) | 41 | 12
Hypophosphataemia (Metabolism and nutrition disorders) | 24 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 31 | 18
Pain in extremity (Musculoskeletal and connective tissue disorders) | 18 | 12
Bone pain (Musculoskeletal and connective tissue disorders) | 15 | 13
Dizziness (Nervous system disorders) | 26 | 16
Rash (Skin and subcutaneous tissue disorders) | 23 | 9
Upper respiratory tract infection (Infections and infestations) | 21 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 52 | 17
Productive cough (Respiratory, thoracic and mediastinal disorders) | 23 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.